CLINICAL TRIAL: NCT04567719
Title: The Role of Bladder Cancer TAS2R38 Expression on Chemotherapy-Induced Bitter Taste
Brief Title: Measuring Taste Perception During Chemotherapy for Muscle Invasive Bladder Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2019-BitterTaste
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Bladder Cancer
Keywords: Musle Invasive
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tongue scrapings will be used for the measurement of TAS2R38 receptor expression by DNA, RNA, and protein.
  Samples from the participant's existing bladder biopsy specimen and radical cystectomy specimen will be obtained and TAS2R38 receptor expression will be measured by DNA, RNA, and protein.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Changes in Taste Perception After Exposure to Chemotherapy: A total of 20 participants with histologically-proven MIBC planning to receive pre-surgery chemotherapy followed by radical cystectomy will be recruited.

SUMMARY:
Alteration in the sense of taste is a frequent symptom that is closely linked to chemotherapy exposure, lowering quality of life and nutritional status. Malnutrition is of particular concern in muscle-invasive bladder cancer (MIBC), as malnutrition is associated with many negative outcomes from radical cystectomy (the surgical procedure in MIBC), which include higher morbidity, poor wound healing, and higher rate of infections after surgery.

It is essential to understand taste changes among participants receiving chemotherapy for MIBC to create future treatment trials.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent.
* Age ≥ 18 years.
* Histologically proven MIBC (Muscle Invasive Bladder Cancer) without metastatic disease Diagnosis.
* Planning to undergo neoadjuvant chemotherapy and radical cystectomy for MIBC

Exclusion Criteria:

* No prior systemic chemotherapy for MIBC.
* Cannot be simultaneously enrolled in any therapeutic clinical trial, unless receiving standard neoadjuvant chemotherapy on said clinical trial.
* Any oral or cognitive pathology impairing the ability to perform taste testing procedures.
* No other known malignancy within previous 2 years with the following EXCEPTIONS: Low-grade prostate cancer on active surveillance, CLL on surveillance / observation, non-melanoma skin cancers.
* No psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from the University Of Kansas Cancer Center.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Perceived strength of taste for the bitter and sweet tastes | From baseline (0-14 days prior to initial chemotherapy) until day of surgery (prior to participant undergoing surgery)
  Taste solution testing using Spectrum(TM) Descriptive Analysis Method. Taste perception is measured on an ordinal scale (e.g. Moderate, Strong, Very Strong).

SECONDARY OUTCOMES:
Changes in nutrition status | 0-14 days prior to initial chemotherapy until (before) day of surgery
  Patient-Generated Subjective Global Assessment (PG-SGA).The PG-SGA Short Form consist of four questions for the participant to rate their weight, food intake, any symptoms they are experiencing and their activity level, with each answer having a numerical correspondence. That score will be combined with the providers health assessment of weight loss, other health conditions that could affect nutrition, any present symptoms and physical exam; again each evaluation will be given a numeric value. The combined scores will determine the participants level of health; with A being well nourished, B being moderate/ suspected malnourished and C being severely malnourished.
Change in body composition | 0-14 days prior to initial chemotherapy until (before) day of surgery
  The Bodystat Quadscan 4000® will measure body fat, lean muscle mass and hydration by placing electrodes on the participants hands and feet. This will show either a resistance or reactance of the electrical flow to determine change in body composition, if any.
TAS2R38 expression in tongue and tumor/ tumor- adjacent tissues | 0-14 days prior to initial chemotherapy until (before) day of surgery
  Tongue scraping and tumor tissue will be collected and tested for TAS2R38 in the DNA, RNA and protein.
Differences between nutrition status at protocol scheduled visits | 0-14 days prior to initial chemotherapy until (before) day of surgery
  Wilcox signed- rank test will compare each score to determine the changes. The scores will be calculated as either positive or negative numbers. If the total score is positive this will indicate that these measurements are related to taste perception. A negative score will show they are not.
Difference between body composition at protocol scheduled visits | 0-14 days prior to initial chemotherapy until (before) day of surgery
  Wilcox signed- rank test will compare each score to determine the changes. The scores will be calculated as either positive or negative numbers. If the total score is positive this will indicate that these measurements are related to taste perception. A negative score will show they are not.
Difference between TAS2R38 expression at protocol scheduled visits. | 0-14 days prior to initial chemotherapy until (before) day of surgery
  Wilcox signed- rank test will compare each score to determine the changes. The scores will be calculated as either positive or negative numbers. If the total score is positive this will indicate that these measurements are related to taste perception. A negative score will show they are not.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Wulff- Burchfield, MD, Principal Investigator — The University of Kansas Cancer Center
Locations (2):
- United States (2):
  - The University of Kansas Medical Center, Kansas City, Kansas
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: No